CLINICAL TRIAL: NCT06049316
Title: Comparative Effects of Scapular Stabilization Versus Scapular Functional Exercises on Chronic Neck Pain.
Brief Title: Scapular Stabilization vs Functional Exercises on Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0135NoorUlHuda
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Neck Pain
Keywords: Neck pain; Scapular exercises; Range of motion; Disability
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scapular stabilization exercises (Experimental): Scapular stabilization exercises
  Interventions: Other: Scapular stabilization exercises
- Scapular functional exercises (Active Comparator): Scapular functional exercises
  Interventions: Other: Scapular functional exercises

INTERVENTIONS:
Other: Scapular stabilization exercises — In Scapular stabilization exercise, following treatment protocol will involve.
  * In supine position, for the relaxation of body, patient will take a deep breath.
  * In sitting position, patient will sit on the chair, placed both feet on the floor while bending knee at 90 degree. After this patient will raise his hand overhead with 90 degree flexion and elbow extension and also perform scapular retraction. (10 sec hold, 10 reps, 20 sec break).
  * In quadrupled position with 120 degree flexion and shoulder abduction patient will lifted his hands. (10 sec hold, 10 reps, 20 sec break) TYI exercises will be administered
  * T shape: Place both arms horizontal with thumbs up. (10 times, 5 sec hold, 3 sets)
  * Y-shape: In prone lying place arms in 45 degree. (10 times, 5 sec hold, 3 sets)
  * I-shape: In prone position patients will place his both arms overhead. (10 times, 5 sec hold, 3 sets).
  These above exercises will perform 3 times a week for eight weeks.
  Arms: Scapular stabilization exercises
Other: Scapular functional exercises — In Scapular functional exercises, following treatment protocol will involve
  * Press-up (in a chair).
  * Push-up plus, Grade 1, in oblique position exercise will be performed with the support of a table. After progression perform this in horizontal plane.
  * Lateral pull down
  * Horizontal pull apart
  * Prone flexion: in prone position on plinth. Both arms placed overhead, and then raise arms towards ceiling.
  * Prone rows: in prone position, with elbow straight, slowly raise arms towards ceiling while bending the elbows.
  These all above exercises will perform by holding dumbbells in hands (20RM at first week, 10RM at last week) with 3 sets, 3 times a week for eight weeks.
  Arms: Scapular functional exercises

SUMMARY:
This project is a Randomized clinical trial, will be conducted to check the comparative effects of scapular stabilization versus scapular functional exercises in patients with chronic neck pain. Study duration will be of 8 months, convenient sampling will be done, subject following eligibility criteria from Amina Physical therapy and rehab Centre Lahore, will be randomly allocated in two groups, baseline assessment will be done, Group A participants will be given baseline treatment along with scapular stabilization exercises, Group B participants will be given baseline treatment along with scapular functional exercises. Assessment will be done in 4th week and 8th week via, Visual analogue scale for neck pain, Function of neck will be assessed by Neck disability index and inclinometer measurements of cervical ranges,3 sessions per week will be given, data will be analyzed by using SPSS version 21.

DETAILED DESCRIPTION:
In recent years musculoskeletal related problems are the leading cause of discomfort in people worldwide. Chronic neck pain is among the most commonly reported problems to physicians. Even before reporting to clinics there is long history of using over the counter pain killers. For the duration of rehabilitation in patients who are suffering from chronic neck pain, exercising has been considered one of the maximum proof-based modalities. Rehabilitation exercises that aim to return functionality of the scapular muscles are deemed necessary to render a successful result on chronic neck pain. In previous researches no one explains the specific treatment protocol in scapular exercises. The current study has compared the effects of scapular stabilization exercises and scapular functional exercises protocol and also compare which is more effective for chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders.(18-35 years of age)
* Patients having chronic neck pain(>3 months duration)
* Patient with restricted ROM of cervical.
* VAS≥4(16)
* NDI ≥10

Exclusion Criteria:

* History of Head, Neck, cervical spine and shoulder injury.
* History of cervical radiculopathy
* History of malignancy, scoliosis, torticollis
* Diagnosed cases of disc prolapse, stenosis, herniation, spondylolisthesis, osteoporosis, and those with current use of any medication or physical therapy treatment were excluded.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
VAS | 8th Week
  This VAS will be used in this study to measure Pain. Patients will be instructed to assess the severity of neck pain experienced last week on a 0-10 cm horizontal line (0 = painless and 10 = worst pain imaginable).
NDI | 8th Week
  NDI will be used to measure function of neck. Neck disability index is the first tool to measure the self-reported disability in patients with neck pain. Total score of NDI is 50 and ranges are defined on the level of disability.
Inclinometer | 8th Week
  Cervical spine range of motion will be assessed by inclinometer. It consists of a circular, fluid-filled disk with a bubble that indicates the number of degrees on the scale of protractor. Bubble inclinometer showed good intrarater and interrater reliability with intraclass Correlation Coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil ur Rehman, Principal Investigator — Riphah International University, Lahore, Pakistan; Noor Ul Huda, Principal Investigator — Riphah International University, Lahore, Pakistan
Locations (1):
- Amina Physical Therapy and Rehab Centre, Lahore, Pakistan, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abichandani D, Ting JTY, Cancino EE, Althobaiti S, Falla D. Measures of neck muscle strength and their measurement properties in adults with chronic neck pain-a systematic review. Syst Rev. 2023 Jan 16;12(1):6. doi: 10.1186/s13643-022-02162-5. PMID 36642710
- [Background] Fatima A, Veqar Z, Zaidi S, Tanwar T. Effects of scapular stabilization and upper limb proprioception as an adjunct to cervical stabilization in chronic neck pain patients: A randomized controlled trial. J Bodyw Mov Ther. 2022 Jan;29:291-301. doi: 10.1016/j.jbmt.2021.10.016. Epub 2021 Nov 1. PMID 35248285
- [Background] Seo YG, Park WH, Lee CS, Kang KC, Min KB, Lee SM, Yoo JC. Is Scapular Stabilization Exercise Effective for Managing Nonspecific Chronic Neck Pain?: A Systematic Review. Asian Spine J. 2020 Feb;14(1):122-129. doi: 10.31616/asj.2019.0055. Epub 2019 Nov 1. PMID 31668049
- [Background] Raju AS, Apparao P, Swamy G, Chaturvadi P, Mounika RG. A comparative study on deep cervical flexors training and neck stabilization exercises in subjects with chronic neck pain. Indian Journal of Physiotherapy & Occupational Therapy. 2019;13(2):1.
- [Background] Celenay ST, Akbayrak T, Kaya DO. A Comparison of the Effects of Stabilization Exercises Plus Manual Therapy to Those of Stabilization Exercises Alone in Patients With Nonspecific Mechanical Neck Pain: A Randomized Clinical Trial. J Orthop Sports Phys Ther. 2016 Feb;46(2):44-55. doi: 10.2519/jospt.2016.5979. Epub 2016 Jan 11. PMID 26755405
- [Background] MAWAD ANW, MOHAMED H, YARA S. Scapular stabilization exercise versus neck stabilization exercise in females with chronic mechanical neck pain. The Medical Journal of Cairo University. 2021;89(December):2729-34.
- [Background] Kang JI, Choi HH, Jeong DK, Choi H, Moon YJ, Park JS. Effect of scapular stabilization exercise on neck alignment and muscle activity in patients with forward head posture. J Phys Ther Sci. 2018 Jun;30(6):804-808. doi: 10.1589/jpts.30.804. Epub 2018 Jun 12. PMID 29950768
- [Background] Attia AMM, Aboelnour NH, Sherif RA, Saafaan KI. Effect of Manual Pressure Release and Scapular Stabilization Exercises on Myofascial Pain Syndrome Following Neck Dissection Surgery. The Egyptian Journal of Hospital Medicine. 2022;89(1):4668-75.
- [Background] Demir O, Atıcı E, Torlak MS. Therapeutic and stabilization exercises after manual therapy in patients with non-specific chronic neck pain: A randomised clinical trial. International Journal of Osteopathic Medicine. 2023;47:100639.
- [Background] Javdaneh N, Ambrozy T, Barati AH, Mozafaripour E, Rydzik L. Focus on the Scapular Region in the Rehabilitation of Chronic Neck Pain Is Effective in Improving the Symptoms: A Randomized Controlled Trial. J Clin Med. 2021 Aug 8;10(16):3495. doi: 10.3390/jcm10163495. PMID 34441791